CLINICAL TRIAL: NCT01572142
Title: Hyposmia, Cholinergic Denervation and Incipient Cognitive Decline in PD
Brief Title: Decrease in Sense of Smell and Associated Cognitive Decline in Parkinson's Disease
Acronym: OLF
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Professor, University of Michigan
Other Study IDs: R01N5070856
Record Dates: First submitted 2012-04-03; First posted 2012-04-06 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson disease; smell; cognitive
MeSH Terms: conditions — Parkinson Disease; Anosmia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson disease group: Subjects with Parkinson disease

SUMMARY:
The overarching goal of this prospective cohort study is to test the hypotheses that greater severity of hyposmia is associated with increased risk of cognitive decline in PD and that worsening hyposmia parallels progressive cholinergic limbic denervation. To achieve the goals of this project, patients with PD without dementia or at-risk of dementia or with dementia will undergo longitudinal olfactory, cognitive and clinical testing for 2-4 years. AChE [11C]PMP or VAchT (vesicular acetylcholine transporter) [F18]-FEOBV PET will be performed both at study entry and at 2-years (± 6 months) follow-up. Brain MRI scans will also be performed at study entry and at 2-years (± 6 months) follow-up. Brain Beta-amyloid PET will be performed at study entry or at 2 years (± 6 months). Annual olfactory testing will be performed to better understand dynamic changes underlying the clinical and PET outcome measures.

DETAILED DESCRIPTION:
Smell functions will be assessed using a test battery of odor identification, odor memory, and odor discrimination tests.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson disease
* Hoehn & Yahr stage 2 and higher, and/or duration of motor disease 5 years or longer
* 50 and older

Exclusion Criteria:

* other disorders which may resemble PD
* subjects with definite dementia
* subjects with unstable or severe medical disorders
* subjects receiving neuroleptic, anticholinergic, or cholinesterase inhibitor drugs
* subjects in whom MRI imaging is contraindicated
* subjects who have received ionizing radiation that would, together with the current project exposures, exceed exposure limits permissible to research volunteers
* pregnant

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Movement Disorders Clinic, Hospital, Primary Care, Community
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2010-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Olfactory testing | Yearly follow up visits

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Bohnen, M.D., Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Universtiy of Michigan Functional Neuroimaging, Cognitive and Mobility Laboratory, Ann Arbor, Michigan, United States